CLINICAL TRIAL: NCT06734507
Title: Laparoscopy Using the Airseal System Versus Standard Insufflation in Cholecystectomy in Children
Brief Title: Laparoscopic Cholecystectomy Using Airseal in Children
Acronym: VBAS
Status: Completed | Type: Observational
Sponsor: Destinval Christelle (Other)
Responsible Party: Sponsor-Investigator, Destinval Christelle, Dr., University Hospital, Clermont-Ferrand
Organization: University Hospital, Clermont-Ferrand (Other)
Other Study IDs: M24DC1109; NCT05848726 (obsolete NCT alias)
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Gall Stones (& [Calculus - Gall Bladder]); Cholecystitis; Pancreatitis Due to Gallstones; Child, Only
Keywords: Laparoscopy; Cholecystectomy; Airseal; Valveless Trocar; Standard Insufflation; Retrospective Study
MeSH Terms: conditions — Gallstones; Cholecystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- A Group: Group of patient who underwent laparoscopic cholecystectomy using Airseal
- S Group: Group of patient who underwent laparoscopic cholecystectomy using a standard insufflator

SUMMARY:
The goal of this observational study is to compare the use of Airseal versus a standard insufflation, in children who underwent laparoscopic cholecystectomy, between January 2021 and December 2022.

The main questions it aims to answer are:

* amount of analgesics consumed postoperatively
* mean digital pain scale

Data are directly extracted from patients medical files.

The investigators will compare the Airseal group (A group) to the Standard insufflation group (S group) to see if the A group consumes significatively less analgesics and are less painful than the S group.

DETAILED DESCRIPTION:
Choosing to enter the A or the S group depends on the surgeon's choice.

Only the surgeon, the anesthetic and the nurses in the operating room know which type of insufflation has been chosen.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged under 18 years old
* Who underwent laparoscopic cholecystectomy
* From January 2021 to December 2022

Exclusion Criteria:

* Patients older than 18 years old

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients adressed to the University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Amount of analgesics consumed | From the end of surgery to the discharge home, up to 20 days
  Number of takings postoperatively
Mean Digital Pain Scale | From the end of surgery to the discharge home, , up to 20 days
  Digital Pain Scale: minimum is 0 out of 10 (which means no pain) and maximum is 10 out of 10 (which means very painful). Higher scores mean worse outcomes.

SECONDARY OUTCOMES:
Operating time | Perioperatively
  Time-length of surgery
Anesthetic time | Perioperatively
  Time-length of anesthesia
Length of stay | From the day of hospitalization to the day of discharge home, up to 20 days
  Hospital length of stay
Histological results | Between 2 weeks and 4 weeks after surgery
  Analysis of the gall bladder after removal

CONTACTS AND LOCATIONS:
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hua J, Gong J, Yao L, Zhou B, Song Z. Low-pressure versus standard-pressure pneumoperitoneum for laparoscopic cholecystectomy: a systematic review and meta-analysis. Am J Surg. 2014 Jul;208(1):143-50. doi: 10.1016/j.amjsurg.2013.09.027. Epub 2014 Jan 16. PMID 24503370
- [Background] de'Angelis N, Petrucciani N, Giannandrea G, Brunetti F. The protocol of low-impact laparoscopic cholecystectomy: the combination of mini-laparoscopy and low-pressure pneumoperitoneum. Updates Surg. 2018 Dec;70(4):553-556. doi: 10.1007/s13304-018-0591-8. Epub 2018 Aug 29. PMID 30159821